CLINICAL TRIAL: NCT03629067
Title: A Randomized, Open-label, Single Dose, 3x3 Partial Replicated Crossover Study to Evaluate the Pharmacokinetics and Safety/Tolerability Between BR1010 and Co-administration of BR1010-1 and BR1010-2 in Healthy Volunteers
Brief Title: Combination of Fimasartan/Amlodipine/Hydrochlorothiazide in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR1010(BR-FAHC-CT-102)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Pharmacokinetics
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence A (Experimental): Period 1(Treatment R) - Period 2(Treatment R) - Period 3(Treatment T)
  There will be a 14 washout of days between the each period.
  Interventions: Drug: Treatment T; Drug: Treatment R
- Sequence B (Experimental): Period 1(Treatment R) - Period 2(Treatment T) - Period 3(Treatment R)
  There will be a 14 washout of days between the each period.
  Interventions: Drug: Treatment T; Drug: Treatment R
- Sequence C (Experimental): Period 1(Treatment T) - Period 2(Treatment R) - Period 3(Treatment R)
  There will be a 14 washout of days between the each period.
  Interventions: Drug: Treatment T; Drug: Treatment R

INTERVENTIONS:
Drug: Treatment T — Fixed dose Combination of Fimasartan/Amlodipine/Hydrochlorothiazide
  Other Names: FAH
Drug: Treatment R — Co-administration of Fimasartan/Amlodipine and Hydrochlorothiazide
  Other Names: FA/H

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetics and safety/tolerability between Fimasartan/Amlodipine/Hydrochlorothiazide and co administration of Fimasartan/Amlodipine and Hydrochlorothiazide in Healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A healthy adults aged 19-50 years

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease
* Hypersensitivity to ingredient of IP and other medication, food
* Participation in any other study within 3months
* History of whole blood donation within 2months and Apheresis 1month

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Cmax | 0~144hours after Medication
  Maximum Concentration of Fimasartan, Amlodipine, Hydrochlorothiazide in plasma

SECONDARY OUTCOMES:
AUCinf | 0~144hours after medication
  "Area under the plasma concentration versus time curve " of Fimasartan, Amlodipine, Hydrochlorothiazide

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea